CLINICAL TRIAL: NCT05990907
Title: Pilot Study: Influence of Ischemic Preconditioning on the Orthostatic Competence of the Microcirculation in the Lower Extremity
Brief Title: Influence of RIC on the Orthostatic Competence of the Microcirculation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISAR Klinikum (Other)
Responsible Party: Principal Investigator, Peter Paul Pfeiler, MD, chief resident, ISAR Klinikum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIC-KIP
Record Dates: First submitted 2023-07-30; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Microcirculation; Orthostatic Intolerance; Remote Ischemic Preconditioning; Hemodynamics
Keywords: Microcirculation; Remote ischemic preconditioning
MeSH Terms: conditions — Orthostatic Intolerance

STUDY DESIGN:
Intervention Model Description: The research project is a controlled, single-arm, monocentric clinical study. Due to the study design, randomization and blinding are not possible.
  Unfortunately, there is no scientific data on how long the effects of ischemic preconditioning last. Thus, in a cross-over design study with protocols 1 and 2 in a different order, there would be a risk or bias that subjects who received ischemic preconditioning in the first measurement would have this effect in the second measurement. For this reason, we decided on a standardized procedure for measurement 1 (without ischemic preconditioning) and measurement 2 (with ischemic preconditioning). In this case, the study design would be one-armed.
Masking Description: Due to the study design, randomization and blinding are not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tilting table without and with RIC (Other): The experimental setup consists of two separate measurements. In the first measurement, the subject is ortho-statically stressed by changing the position (lying to upright) on a tilting table (similar to the established tilting table test). 24 hours after the first measurement, the ischemic preconditioning will be carried out in three cycles with a directly subsequent tilting table test.
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — The empty tourniquet (VBM Tourniquet Touch®, Sulz a.N. Germany) is attached to the right upper arm. The measurement starts from this point in time. After lying flat for 10 minutes, the upper arm tourniquet is inflated to 250 mmHg. In all subjects, the ischemia was verified by palpation and Doppler signal of the radial artery. The ischemia phase is carried out for 10 minutes, so the tourniquet is opened and a 10-minute reperfusion phase is started, followed by a total of 3 cycles. After the 3rd ischemia phase, the tilting table test is followed by a 15-minute lying interval.

SUMMARY:
The goal of this clinical trial (pilot study) is to learn about the microcirculatory regulation of the lower extremity under orthostatic stress with and without RIC - Remote Ischemic Preconditioning in healthy participants. The main question it aims to answer are:

Do the beneficial effects of RIC withstand orthostatic stress? / Does RIC benefit lower extremity microcirculation in ortho-statically stressed subjects? Is there a relationship/correlation between the variables of microcirculation and hemodynamics in the context of RIC and orthostatic loading?

DETAILED DESCRIPTION:
The use of free flaps is a standard procedure in reconstructive plastic surgery, in which a wide variety of tissue units are microsurgically transplanted, often to cover defects on the body surface. Microvascular tissue transplants depend on an adequate blood supply, which is particularly vulnerable in the first postoperative phase. In the case of reconstructions of the lower extremities in particular, the flap perfusion is stressed during the first mobilizations due to the orthostatic load. For this reason, the mobilization of the patients is gradually increased from day to day with precise monitoring of the blood flow (so-called flap training).

A procedure for temporarily improving the blood flow in free flaps is ischemic preconditioning (RIC - Remote Ischemic Preconditioning). Repeated, short cycles of ischemia/reperfusion applied to a circumscribed vascular territory (e.g. supra systolic tourniquet arm) lead to an increase in tissue perfusion, even outside the area of application (arm).

RIC could have the potential to optimize the tissue perfusion of flaps even under orthostatic stress and to promote an earlier mobilization of patients. Our work investigates the influence of RIC on orthostatic competence (as part of a standardized orthostatic load with a tilting table) of the microcirculatory system in the lower extremities and the orthostatic hemodynamic regulation itself.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* No diseases relevant to circulation and blood flow (arterial hypertension, peripheral arterial occlusive disease, chronic venous insufficiency)
* Subjects must be capable of insight. Anyone who can understand the nature, significance, and scope of the clinical trial and determine their will accordingly is capable of insight.

Exclusion Criteria:

* Non-consent
* Lack of compliance
* Syncope tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-08-13 (Estimated)

PRIMARY OUTCOMES:
Microcirculation parameters | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  Microcirculation parameter (Measured with O2C laser Doppler and tissue spectrometry LEA Medizintechnik GmbH, Giessen, Germany) Relative blood flow in arbitrary units [AU]

SECONDARY OUTCOMES:
Microcirculation parameters - oxygen saturation | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  Microcirculation parameter (Measured with O2C laser Doppler and tissue spectrometry LEA Medizintechnik GmbH, Giessen, Germany) capillary venous oxygen saturation in percent (%)
Microcirculation parameters - Relative amount of hemoglobin | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  Microcirculation parameter (Measured with O2C laser Doppler and tissue spectrometry LEA Medizintechnik GmbH, Giessen, Germany) Relative amount of hemoglobin in arbitrary units [AU]
Hemodynamics | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  hemodynamics parameters: systolic blood pressure in mmHg (Measured with Finapres® NOVA, Finapres Medical Systems BV, Enschede, Netherlands)
Hemodynamics | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  hemodynamics parameters: mean arterial blood pressure in mmHg (Measured with Finapres® NOVA, Finapres Medical Systems BV, Enschede, Netherlands)
Hemodynamics | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  hemodynamics parameters: diastolic blood pressure in mmHg (Measured with Finapres® NOVA, Finapres Medical Systems BV, Enschede, Netherlands)
Hemodynamics | continuous measurement; Focus on the following periods: 1 minute before RIC, 1 min before the tilting table, half-time minute in the upright position, 1 min before the end of the measurment
  hemodynamics parameters: heart rate in beats per minute (Measured with Finapres® NOVA, Finapres Medical Systems BV, Enschede, Netherlands)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, MD, PhD, Study Chair — Department Plastic Surgery ISAR Klinikum, Munich
Locations (1):
- ISAR Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT05990907/Prot_000.pdf